CLINICAL TRIAL: NCT03543748
Title: Efficacy and Safety of rTMS for Cognitive Rehabilitation in Moyamoya Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yu Lei, attending doctor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ylei
Record Dates: First submitted 2017-12-15; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-04

CONDITIONS: Moyamoya Disease
Keywords: Transcranial Magnetic Stimulation; cognitive impairment
MeSH Terms: conditions — Moyamoya Disease; Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TMS (Experimental): The Transcranial Magnetic Stimulation course consisted of daily sessions of 2,000 stimuli for the left DLPFC (50 trains of 40 stimuli at 10 Hz for 10 days),
  Interventions: Device: Transcranial Magnetic Stimulation
- SHAM (Sham Comparator): The patient is treated with Sham-TMS stimulation according to protocol with an inactive coil. The sham coil looks and sounds just like the real coil, but produces a negligible magnetic field.
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — A total of 2000 trains will be delivered successively. The pulses will be delivered at 80% of motor thresholds.
  Other Names: TMS
  Arms: TMS
Device: Sham Transcranial Magnetic Stimulation — The sham coil looks and sounds just like the real coil, but produces a negligible magnetic field.
  Other Names: Sham-TMS
  Arms: SHAM

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of transcranial magnetic stimulation (TMS) therapy in moyamoya patients who received surgical revascularization.

DETAILED DESCRIPTION:
Primary Outcome Measures:

TMS stimulation applied to the left DLPFC has a quantifiable effect on cognition [ Time Frame: Neuropsychological Assessments: Baseline（7days after STA-MCA bypass surgery）; 2 months after TMS treatment Changes in one or more assessed cognitive domains at baseline will be measured by comparing the scores for the different neuropsychological tests.

Secondary Outcome Measures:

Change in structural grey and white matter in the brain at baseline compared to after TMS stimulation [ Time Frame: MRI: Baseline and two months after TMS stimulation ] MRI analysis will measure any changes in cortical thickness (mm) or other structural changes in the brain after TMS or Sham-TMS stimulation

Change in executive functioning measured as resting-state functional MRI (fMRI) sequence [ Time Frame: MRI: Baseline and two months after TMS stimulation ] fMRI analysis will measure any changes in amplitude of low frequency fluctuation(ALFF) and other functional changes after TMS stimulation compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. right-handed Chinese population aged 18-80 years;
2. No evidence of infarct in the cerebral cortex, basal ganglia, brainstem, or cerebellum, but small patches of hyper intense signal neither larger than the arbitrary cut off of 8 mm in maximum dimension on T2-weighted MR images no cystic in the cerebral subcortical white matter could be involved;
3. No evidence of intracerebral hemorrhage;
4. diagnosis through digital subtraction angiography;
5. physically capable of cognitive evaluation;
6. absence of significant psychiatric disorders or neurological diseases;
7. No evidence of perioperative epilepsy.

Exclusion Criteria:

1. Significant neurological diseases or psychiatric disorders that could affect cognition
2. Other cerebrovascular diseases (such as atherosclerosis or vasculitides) likely to cause focal cerebral ischemia
3. Concomitant cerebrovascular diseases (such as aneurysms or arteriovenous malformation) that need surgical intervention
4. Severe systemic diseases pregnant or perinatal stage women
5. Any diseases likely to death within 2 years
6. Taking drugs such as benzodiazepine clonazepam
7. Allergy to iodine or radiographic contrast media
8. Concurrent participation in any other experimental treatment trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive outcomes at 3 months follow-up after TMS | 3 months
  Measure neurocognitive outcomes using Mini-mental State Examination (MMSE)
Neurocognitive outcomes at 3 months follow-up after TMS | 3 months
  Measure neurocognitive outcomes using memory and executive screening (MES)

SECONDARY OUTCOMES:
Change in structural imaging in the brain at baseline compared to after TMS stimulation | 3 months
  MRI analysis will measure any changes in cortical thickness (mm) in the brain after TMS or Sham-TMS stimulation
Change in structural imaging in the brain at baseline compared to after TMS stimulation | 3 months
  MRI analysis will measure any changes in cortical white matter micro-structure (DTI) in the brain after TMS or Sham-TMS stimulation
Change in functional imaging in the brain at baseline compaired to after TMS stimulation | 3 month
  MRI analysis will measure any changes in ALFF in the brain after TMS or Sham-TMS stimulation
Change in functional imaging in the brain at baseline compaired to after TMS stimulation | 3 month
  MRI analysis will measure any changes in functional connectivity strength in the brain after TMS or Sham-TMS stimulation